CLINICAL TRIAL: NCT00609843
Title: Lipiodol Demarcation of the Bladder Tumour in Adaptive Image-guided Radiotherapy: A Pilot Study. (Danish: Lipiodol Til Markering af blæretumoren i Forbindelse Med Adaptiv Billedvejledt strålebehandling: Et Pilotstudie.)
Brief Title: Pilot Studie of Lipiodol Demarcation of the Tumour in Bladder Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PilotBladder-IGRT
Record Dates: First submitted 2008-01-24; First posted 2008-02-07 (Estimated); Last update posted 2015-12-07 (Estimated); Status verified 2009-07

CONDITIONS: Bladder Cancer
Keywords: Bladder cancer; Radiotherapy; Tumour delineation; Markers
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental)
  Interventions: Other: Lipiodol demarcation of the bladder tumour

INTERVENTIONS:
Other: Lipiodol demarcation of the bladder tumour — 1-3 drops of Lipiodol Ultra Fluid (iodine 38%W/W) will be injected into the submucosa on 4 locations around the bladder tumour. The procedure is done once during a planned cystoscopy approximately a week before the planning CT.

SUMMARY:
Rationale: Bladder tumours are often not visible on X-ray based image-modalities during planning and treatment of Radiotherapy.

Purpose: To determine if a single contrast (Lipiodol) demarcation of the bladder tumour before treatment is feasible and visible on multiple X-ray based image-modalities during Radiotherapy.

DETAILED DESCRIPTION:
To exploit the potential of modern Radiotherapy (RT), it is important to localize and follow the target precisely during treatment. Since the bladder tumour can usually not be identified on conventional CT-scan, a fiducial or contrast marking system is warranted.

The iodized oil, Lipiodol is a well-known contrast media used mainly for lymphography and Hysterosalpingography. Local Lipiodol demarcation has been used for localisation of tumours in the lung, prostate and seminal vesicles visualised on Computed Tomography (CT) and fluoroscopy.

Purpose: To evaluate the feasibility of tumour demarcation using the contrast agent Lipiodol in adaptive Image-guided RT of bladder cancer. Visibility on CT, Cone-Beam CT, MRI and on-board imaging will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed primary muscle invasive transitional cell carcinoma of the Bladder. T1-4a, N0-1, M0.
* Non-operable or refuse operation.
* Eligible for curative Radiotherapy.
* Oral and written informed consent.
* Fertile women must have a negative pregnancy test before inclusion or use contraceptive pills or intrauterine device.
* Ongoing beta blocker treatment is paused before Lipiodol injection.

Exclusion Criteria:

* Known metabolic disorder (hyperthyroidism, goiter)
* Allergy towards iodine.
* Pregnancy / breast-feeding
* Performance status ECOG > 2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2008-02; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Is Lipiodol demarcation visible on the planning CT (Feasibility) | Before Radiotherapy
Is Lipiodol visible on CBCT during Radiotherapy treatment (duration) | Daily the first week, then two times a week during Radiotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Jimmi Søndergaard, M.D, Principal Investigator — The Oncologic department of Aarhus Sygehus, Aarhus University Hospital
Locations (1):
- The Oncology department of Aarhus Sygehus, Aarhus University Hospital, Aarhus, Central Jutland, Denmark

REFERENCES:
- [Derived] Sondergaard J, Olsen KO, Muren LP, Elstrom UV, Grau C, Hoyer M. A study of image-guided radiotherapy of bladder cancer based on lipiodol injection in the bladder wall. Acta Oncol. 2010 Oct;49(7):1109-15. doi: 10.3109/02841861003789491. PMID 20429726